CLINICAL TRIAL: NCT06127004
Title: Metacognitive Training for Negative Symptoms (MCT Minus)
Brief Title: Metacognitive Training for Negative Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sormland County Council, Sweden (Other)
Collaborators: Uppsala County Council, Sweden (Other Government); Västmanland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Region Sörmland; Department of Medical Sciences (Other: Uppsala Univsersity)
Record Dates: First submitted 2023-07-22; First posted 2023-11-13 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Negative Symptoms in Schizophrenia

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metacognitive Training for Negative Symptoms (Experimental): The original MCT intervention was adapted to negative symptoms by incorporating psychoeducation and strategies to target the cognitions suggested by the cognitive model (Beck et al., 2009) to be implicated in the development and/or maintenance of negative symptoms. Although some of the strategies have traditionally been used to target positive symptoms, it is assumed that the same reasoning styles lead to negative symptoms through the dysfunctional cognitions discussed previously (e.g., jumping to conclusions in regard to social rejection and a dysfunctional attribution style reinforcing social withdrawal). Metacognitive training for negative symptoms consists of eight sessions, delivered individually as there is evidence indicating that this approach may lead to stronger effect sizes than delivery in a group format (Liu et al., 2018). The developer of MCT (Professor Steffen Moritz) approved the modification.
  Interventions: Other: Metacognitive Training for Negative Symptoms (MCT)
- Control group (Active Comparator): Supportive Counselling (8 sessions) will be used as a control. Participants enrolled in this condition can then get the intervention if they request this.
  Interventions: Other: Supportive Counselling

INTERVENTIONS:
Other: Metacognitive Training for Negative Symptoms (MCT) — See arm/group descriptions
  Arms: Metacognitive Training for Negative Symptoms
Other: Supportive Counselling — Se arm/group descriptions
  Arms: Control group

SUMMARY:
There is a clear rationale for developing interventions targeting negative symptoms of schizophrenia as these are a stronger indicator of current and future functioning than positive symptoms and because they respond poorly to medication and existing psychological interventions. This is reflected in the NIMH-MATRICS consensus statement that emphasised that persistent negative symptoms represent an unmet therapeutic need for patients suffering from schizophrenia.

The purpose of this study is to evaluate, in a scientific manner, the intervention developed by Swanson et al. 2021: Metacognitive Training (MCT) Minus. The MCT was adapted to target negative symptoms in psychotic disorders (e.g. schizophrenia, schizoaffective or non-affective functional psychosis) as the original version of the intervention focused exclusively on positive symptoms. The specific aim is to study whether MCT Minus is a promising treatment for the intended population in terms of reductions in negative symptoms, severity of defeatist attitudes, internalised stigma, and depression as well as improvements in reflective ability and overall functioning.

The research will add to existing research by identifying and measuring potential mechanisms of change for negative symptoms (i.e., defeatist attitudes, reflective functioning, stigma and depression). It will also add to the existing evidence base by measuring whether the cognitive biases addressed in MCT lead to changes in the wider conceptualisation of metacognition used elsewhere and whether the promising results seen in the feasibility study of MCT Minus can be replicated in a randomised controlled trial (RCT) with a control group and a blinded assessor. The researchers also hope to replicate the findings of a previous study, where MCT was found to be related to the modulation of default-mode network (DMN) homogeneity in schizophrenia, an area thought to be involved in self- and other-reflectivity.

DETAILED DESCRIPTION:
Introduction:

While clinicians tend to focus on positive symptoms as primary treatment targets in schizophrenia, patients prioritize the treatment of depressive and negative symptoms. Persistent negative symptoms are experienced by approximately 20%-40% of individuals diagnosed with schizophrenia. Current research indicates that negative symptoms are independent from positive symptoms, depression, cognitive dysfunctions, and disorganization. However, neither medication nor existing psychosocial interventions have proven to be efficacious in reducing negative symptoms. Consequently, authors have highlighted the need for better understanding of treatment mechanisms underpinning psychological interventions that directly target negative symptoms.

Psychological conceptualizations suggest that negative symptom expression can, in some cases, be understood as a response to adverse experiences. For example, Beck et al.'s cognitive model suggests that negative symptoms emerge from a process where individuals adopt coping strategies of 'shutting down' the cognitive-affective experience. This allows individuals to cope with overwhelming or aversive situations in the short term but leads to a reliance on negative symptoms (including social withdrawal, avolition, and diminished expression) to reduce exposure to, and impact of, negative experiences in the longer term. From an attachment framework, Griffiths and McLeod (2019) suggest that negative symptoms may be seen 'as responses involving emotional and social withdrawal that emerge from threats to self-security'. If negative symptoms can be understood within cognitive and developmental frameworks, it may be possible to develop theoretically driven interventions for their treatment.

A cognitive model of negative symptoms:

Negative symptoms are associated with low expectations of future success, asocial beliefs, a reduced sense of self-efficacy, negative self-concepts, defeatist performance beliefs and self-stigma. The cognitive model therefore proposes that negative symptoms might be caused and maintained by dysfunctional beliefs arising as a consequence of repeated failures and setbacks. These appraisals might include negative beliefs about social affiliations; low expectations of pleasure, success and acceptance; defeatist beliefs about performance; and a perception of limited resources. The self-perception, and perceived self-efficacy, of individuals diagnosed with schizophrenia may also be influenced by self-stigmatizing views of their mental illness. It might be that these factors result in hypervigilance to perceived criticism. Longitudinal studies have shown support for the cognitive model as defeatist performance attitudes and asocial beliefs are found to predict future negative symptoms.

Metacognition and psychosis:

Metacognition was initially referred to as the capacity to think about and monitor one's mental processes. However, the definition has broadened in contemporary research, ranging 'from discrete processes involving noticing specific thoughts and feelings to more synthetic acts in which information is integrated into complex representations of the self and others'. This has given rise to interventions targeting metacognitive processes, some of which have been specifically developed for psychosis e.g., metacognitive training (MCT); metacognitive reflection and insight therapy (MERIT), while others have been modified for this population. MCT is based on the premise that cognitive biases play a role in the development and maintenance of psychotic symptoms which can be alleviated by targeting underlying cognitive processes. The aims are to gain insight and to learn practical strategies to manage distressing symptoms. MCT has been shown to reduce delusions and positive symptoms and improve cognitive insight and biases. Preliminary evidence also suggests effects on quality of life and illness insight.

Several authors highlight the links between negative symptoms and compromised capacity for self/others mental state processing. There is evidence that suggests a link between metacognition and negative symptoms as limitations in complex metacognitive processes predict negative symptoms in first episode psychosis and in more chronic samples, even after controlling for defeatist beliefs, affect recognition and neurocognitive functioning. Metacognitive deficits are also associated with concurrent and future negative symptoms when controlling for verbal memory and education. Interestingly, self-reflection in itself has been found to mediate the relationship between neurocognition and negative symptoms (especially for deficits in capacity to communicate about internal states, so called diminished expression) while interpersonal cognitive differentiation (i.e., the ability to construe one's experiences as either similar or different from others' experiences) has been found to mediate the pathway between self-reflectivity and negative symptoms. This suggests that negative symptom reduction may at least partially depend on improved metacognitive capacity and that a metacognitive intervention specifically targeting negative symptoms may be beneficial.

Swanson et al. (2021) therefore adapted MCT for negative symptoms to assess the acceptability and feasibility of the intervention, examine variable change over the course of the intervention and carry out a preliminary investigation of putative mechanisms of change. The current project is a further evaluation of this, where the researchers hope to achieve similarly encouraging results in a randomised controlled trial (RCT) with a control group and blinding. The researchers also hope to replicate the findings of a previous study where MCT was found to be related to the modulation of default-mode network (DMN) homogeneity in schizophrenia, an area thought to be involved in self- and other-reflectivity. Importantly, it was found that high network homogeneity levels at baseline in the bilateral superior medial prefrontal cortex could predict symptomatic improvement after 8 weeks of drug plus psychotherapy treatment; this illustrates that a more developed understanding of the biological mechanisms underlying negative symptoms would allow us to identify patients that would benefit from each type of treatment and, through that, change the prognosis and treatment outcomes of the condition.

Significance and scientific novelty:

Research funding has been given for a RCT to evaluate the intervention trialled by Swanson et al, 2021 in a more rigorous and scientific manner. Given our limited understanding of negative symptoms and how to treat them, the study would be of both significance and scientific novelty. To fully understand the biological mechanisms behind negative symptoms is essential to be able to develop future treatment options and to identify patients that would benefit from each type of treatment. A more thorough understanding of schizophrenia would decrease the heterogeneity of the condition which would have vast implications for how individuals diagnosed with schizophrenia are treated both in society and in the healthcare setting.

Previous results:

Two articles (which were based on the main researcher's doctoral thesis at Edinburgh University with funding from National Health Service (NHS) Lothian) have been published in Clinical Psychology and Psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Clinical diagnosis of schizophrenia, delusional disorder or non-affective psychosis
* Resident in Region Sörmland, Region Västmanland or Region Uppland

Exclusion Criteria:

* Evidence of severe organic brain dysfunction
* Learning disabilities
* Difficulty with the Swedish language
* Visual and/or hearing impairment
* Being unable or unwilling to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
The Clinical Assessment Interview for Negative Symptoms (CAINS) (Forbes et al., 2011) | 15 minutes
  Clincial interview to assess negative symptoms.
  Minimum value is 0 = better outcome. Maximum value is 52 = worse outcome.
The Motivation and Pleasure Scale- Self-Report (MAP-SR) (Llerena et al., 2013) | 5 minutes
  Self-rated questionnaire to assess negative symptoms
  Minimum value is 0 = better outcome. Maximum value is 90 = worse outcome.
The Positive and Negative Syndrome Scale (PANSS) (Kay et al., 1987) | 20 minutes
  Clinical interview to assess negative symptoms (analysed with the five factor-model)
  Minimum value is 0 = better outcome. Maximum value is 210 = worse outcome.

SECONDARY OUTCOMES:
The Dysfunctional Attitudes Scale (DAS) (Weissman & Beck, 1978) | 5 minutes
  Self-rated questionnaire to assess defeatist attitudes
  Minimum value is 100 = better outcome. Maximum value is 700 = worse outcome.
The Reflective Functioning Questionnaire (RFQ-8) (Fonagy et al., 2016) | 5 minutes
  Self-rated questionnaire to assess metacognitive ability
  Minimum value is 8 = worse outcome. Maximum value is 24 = better outcome.
The Internalized Stigma of Mental Illness Scale-9 (ISMI-9) (Hammer & Toland, 2017) | 5 minutes
  Self-rated questionnaire to assess stigma
  Minimum value is 1 = better outcome. Maximum value is 4 = worse outcome.
The Calgary Depression Scale for Schizophrenia (CDSS) (Addington, Addington, & Schissel, 1990) | 10 minutes
  Clinical interview to assess depressive symptoms in schizophrenia
  Minimum value is 0 = better outcome. Maximum value is 36 = worse outcome.
The World Health Organization (WHO) Disability Assessment Schedule (WHODAS) 2.0 (WHO, 2010) | 10 minutes
  Clinical interview to assess overall functioning
  Minimum value is 0 = better outcome. Maximum value is 144 = worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Swanson, Dr, Principal Investigator — Region Sörmland/ Uppsala University
Locations (1):
- Region Sörmland, Multiple Locations, Sweden

IPD SHARING:
Plan to Share IPD: No
Data can be shared on request with other researchers

REFERENCES:
- [Background] Addington D, Addington J, Schissel B. A depression rating scale for schizophrenics. Schizophr Res. 1990 Jul-Aug;3(4):247-51. doi: 10.1016/0920-9964(90)90005-r. PMID 2278986
- [Background] Aleman A, Lincoln TM, Bruggeman R, Melle I, Arends J, Arango C, Knegtering H. Treatment of negative symptoms: Where do we stand, and where do we go? Schizophr Res. 2017 Aug;186:55-62. doi: 10.1016/j.schres.2016.05.015. Epub 2016 Jun 9. PMID 27293137
- [Background] American Psychiatric Association (APA). (1987). Diagnostic and statistical manual of mental disorders (3rd edition, revised) (DSM-III-TR). APA.
- [Background] Austin, S. F., Lysaker, P. H., Jansen, J. E., Trauelsen, A. M., Nielsen, H.-G. L., Pedersen, M. B., Haahr, U. H., & Simonsen, E. (2019). Metacognitive capacity and negative symptoms in first episode psychosis: Evidence of a prospective relationship over a 3-year follow-up. Journal of Experimental Psychopathology, 10(1). doi: 10.1177/2043808718821572
- [Background] Beck, A. T., Rector, N. A., Stolar, N., & Grant, P. (2009). Schizophrenia: cognitive theory, research and therapy. Guilford Press.
- [Background] Beck AT, Himelstein R, Grant PM. In and out of schizophrenia: Activation and deactivation of the negative and positive schemas. Schizophr Res. 2019 Jan;203:55-61. doi: 10.1016/j.schres.2017.10.046. Epub 2017 Nov 21. PMID 29169775
- [Background] Bentall, R. P., Simpson, P. W., Lee, D. A., Williams, S., Elves, S., Brabbins, C., & Morrison, A. P. (2010). Motivation and avolition in schizophrenia patients: The role of self-efficacy. Psychosis, 2(1), 12-22. doi: 10.1080/17522430903505966
- [Background] Birules I, Lopez-Carrilero R, Cuadras D, Pousa E, Barrigon ML, Barajas A, Lorente-Rovira E, Gonzalez-Higueras F, Grasa E, Ruiz-Delgado I, Cid J, de Apraiz A, Montserrat R, Pelaez T, Moritz S, The Spanish Metacognition Study Group, Ochoa S. Cognitive Insight in First-Episode Psychosis: Changes during Metacognitive Training. J Pers Med. 2020 Nov 27;10(4):253. doi: 10.3390/jpm10040253. PMID 33260823
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3(2), 77-101. doi: 10.1191/1478088706qp063oa
- [Background] Campellone TR, Sanchez AH, Kring AM. Defeatist Performance Beliefs, Negative Symptoms, and Functional Outcome in Schizophrenia: A Meta-analytic Review. Schizophr Bull. 2016 Nov;42(6):1343-1352. doi: 10.1093/schbul/sbw026. Epub 2016 Mar 15. PMID 26980144
- [Background] Correll CU, Schooler NR. Negative Symptoms in Schizophrenia: A Review and Clinical Guide for Recognition, Assessment, and Treatment. Neuropsychiatr Dis Treat. 2020 Feb 21;16:519-534. doi: 10.2147/NDT.S225643. eCollection 2020. PMID 32110026
- [Background] Cox C, Jolley S, Johns L. Understanding and treating amotivation in people with psychosis: An experimental study of the role of guided imagery. Psychiatry Res. 2016 Dec 30;246:387-391. doi: 10.1016/j.psychres.2016.09.047. Epub 2016 Sep 28. PMID 27788457
- [Background] Faith LA, Lecomte T, Corbiere M, Francoeur A, Hache-Labelle C, Lysaker PH. Metacognition Is Uniquely Related to Concurrent and Prospective Assessments of Negative Symptoms Independent of Verbal Memory in Serious Mental Illness. J Nerv Ment Dis. 2020 Nov;208(11):837-842. doi: 10.1097/NMD.0000000000001219. PMID 32740145
- [Background] Flavell, J. H. (1979). Metacognition and cognitive monitoring: A new area of cognitive-developmental inquiry. American Psychologist, 34(10), 906-911. doi: 10.1037/0003-066X.34.10.906
- [Background] Fonagy P, Luyten P, Moulton-Perkins A, Lee YW, Warren F, Howard S, Ghinai R, Fearon P, Lowyck B. Development and Validation of a Self-Report Measure of Mentalizing: The Reflective Functioning Questionnaire. PLoS One. 2016 Jul 8;11(7):e0158678. doi: 10.1371/journal.pone.0158678. eCollection 2016. PMID 27392018
- [Background] Forbes C, Blanchard JJ, Bennett M, Horan WP, Kring A, Gur R. Initial development and preliminary validation of a new negative symptom measure: the Clinical Assessment Interview for Negative Symptoms (CAINS). Schizophr Res. 2010 Dec;124(1-3):36-42. doi: 10.1016/j.schres.2010.08.039. Epub 2010 Sep 24. PMID 20869848
- [Background] Fox-Wasylyshyn SM, El-Masri MM. Handling missing data in self-report measures. Res Nurs Health. 2005 Dec;28(6):488-95. doi: 10.1002/nur.20100. PMID 16287052
- [Background] Fusar-Poli P, Papanastasiou E, Stahl D, Rocchetti M, Carpenter W, Shergill S, McGuire P. Treatments of Negative Symptoms in Schizophrenia: Meta-Analysis of 168 Randomized Placebo-Controlled Trials. Schizophr Bull. 2015 Jul;41(4):892-9. doi: 10.1093/schbul/sbu170. Epub 2014 Dec 20. PMID 25528757
- [Background] Galderisi S, Mucci A, Buchanan RW, Arango C. Negative symptoms of schizophrenia: new developments and unanswered research questions. Lancet Psychiatry. 2018 Aug;5(8):664-677. doi: 10.1016/S2215-0366(18)30050-6. Epub 2018 Mar 27. PMID 29602739
- [Background] Galderisi S, Mucci A, Dollfus S, Nordentoft M, Falkai P, Kaiser S, Giordano GM, Vandevelde A, Nielsen MO, Glenthoj LB, Sabe M, Pezzella P, Bitter I, Gaebel W. EPA guidance on assessment of negative symptoms in schizophrenia. Eur Psychiatry. 2021 Feb 18;64(1):e23. doi: 10.1192/j.eurpsy.2021.11. PMID 33597064
- [Background] Garcia-Mieres H, Lundin NB, Minor KS, Dimaggio G, Popolo R, Cheli S, Lysaker PH. A cognitive model of diminished expression in schizophrenia: The interface of metacognition, cognitive symptoms and language disturbances. J Psychiatr Res. 2020 Dec;131:169-176. doi: 10.1016/j.jpsychires.2020.09.008. Epub 2020 Sep 14. PMID 32979692
- [Background] Garcia-Mieres H, Nino-Robles N, Ochoa S, Feixas G. Exploring identity and personal meanings in psychosis using the repertory grid technique: A systematic review. Clin Psychol Psychother. 2019 Nov;26(6):717-733. doi: 10.1002/cpp.2394. Epub 2019 Aug 26. PMID 31412423
- [Background] Granholm E, Holden J, Worley M. Improvement in Negative Symptoms and Functioning in Cognitive-Behavioral Social Skills Training for Schizophrenia: Mediation by Defeatist Performance Attitudes and Asocial Beliefs. Schizophr Bull. 2018 Apr 6;44(3):653-661. doi: 10.1093/schbul/sbx099. PMID 29036391
- [Background] Grant PM, Beck AT. Defeatist beliefs as a mediator of cognitive impairment, negative symptoms, and functioning in schizophrenia. Schizophr Bull. 2009 Jul;35(4):798-806. doi: 10.1093/schbul/sbn008. Epub 2008 Feb 27. PMID 18308717
- [Background] Griffiths, H., & McLeod, H. (2019). Promoting recovery from negative symptoms: An attachment theory perspective. In K. Berry, S. Bucci, & A. N. Danquah (Eds.), Attachment theory and psychosis: Current perspectives and future directions (pp. 62-83). Routledge/Taylor & Francis Group.
- [Background] Gspandl S, Peirson RP, Nahhas RW, Skale TG, Lehrer DS. Comparing Global Assessment of Functioning (GAF) and World Health Organization Disability Assessment Schedule (WHODAS) 2.0 in schizophrenia. Psychiatry Res. 2018 Jan;259:251-253. doi: 10.1016/j.psychres.2017.10.033. Epub 2017 Nov 5. PMID 29091824
- [Background] Gumley AI, Taylor HE, Schwannauer M, MacBeth A. A systematic review of attachment and psychosis: measurement, construct validity and outcomes. Acta Psychiatr Scand. 2014 Apr;129(4):257-74. doi: 10.1111/acps.12172. Epub 2013 Jul 3. PMID 23834647
- [Background] Hammer, J. H., & Toland, M. D. (2017). Internal structure and reliability of the Internalized Stigma of Mental Illness Scale (ISMI-29) and Brief Versions (ISMI-10, ISMI-9) among Americans with depression. Stigma and Health, 2(3), 159-174. doi: 10.1037/sah0000049
- [Background] Harder S. Attachment in schizophrenia--implications for research, prevention, and treatment. Schizophr Bull. 2014 Nov;40(6):1189-93. doi: 10.1093/schbul/sbu133. Epub 2014 Sep 16. PMID 25232144
- [Background] Horsselenberg EM, van Busschbach JT, Aleman A, Pijnenborg GH. Self-Stigma and Its Relationship with Victimization, Psychotic Symptoms and Self-Esteem among People with Schizophrenia Spectrum Disorders. PLoS One. 2016 Oct 26;11(10):e0149763. doi: 10.1371/journal.pone.0149763. eCollection 2016. PMID 27783677
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Kirkpatrick B, Strauss GP, Nguyen L, Fischer BA, Daniel DG, Cienfuegos A, Marder SR. The brief negative symptom scale: psychometric properties. Schizophr Bull. 2011 Mar;37(2):300-5. doi: 10.1093/schbul/sbq059. Epub 2010 Jun 17. PMID 20558531
- [Background] Kumari S, Malik M, Florival C, Manalai P, Sonje S. An Assessment of Five (PANSS, SAPS, SANS, NSA-16, CGI-SCH) commonly used Symptoms Rating Scales in Schizophrenia and Comparison to Newer Scales (CAINS, BNSS). J Addict Res Ther. 2017;8(3):324. doi: 10.4172/2155-6105.1000324. Epub 2017 May 11. PMID 29430333
- [Background] Lincoln TM, Mehl S, Kesting ML, Rief W. Negative symptoms and social cognition: identifying targets for psychological interventions. Schizophr Bull. 2011 Sep;37 Suppl 2(Suppl 2):S23-32. doi: 10.1093/schbul/sbr066. PMID 21860044
- [Background] Liu YC, Tang CC, Hung TT, Tsai PC, Lin MF. The Efficacy of Metacognitive Training for Delusions in Patients With Schizophrenia: A Meta-Analysis of Randomized Controlled Trials Informs Evidence-Based Practice. Worldviews Evid Based Nurs. 2018 Apr;15(2):130-139. doi: 10.1111/wvn.12282. Epub 2018 Feb 28. PMID 29489070
- [Background] Llerena K, Park SG, McCarthy JM, Couture SM, Bennett ME, Blanchard JJ. The Motivation and Pleasure Scale-Self-Report (MAP-SR): reliability and validity of a self-report measure of negative symptoms. Compr Psychiatry. 2013 Jul;54(5):568-74. doi: 10.1016/j.comppsych.2012.12.001. Epub 2013 Jan 22. PMID 23351831
- [Background] Lopez-Morinigo JD, Ajnakina O, Martinez AS, Escobedo-Aedo PJ, Ruiz-Ruano VG, Sanchez-Alonso S, Mata-Iturralde L, Munoz-Lorenzo L, Ochoa S, Baca-Garcia E, David AS. Can metacognitive interventions improve insight in schizophrenia spectrum disorders? A systematic review and meta-analysis. Psychol Med. 2020 Oct;50(14):2289-2301. doi: 10.1017/S0033291720003384. Epub 2020 Oct 14. PMID 33050956
- [Background] Lutgens D, Gariepy G, Malla A. Psychological and psychosocial interventions for negative symptoms in psychosis: systematic review and meta-analysis. Br J Psychiatry. 2017 May;210(5):324-332. doi: 10.1192/bjp.bp.116.197103. Epub 2017 Mar 16. PMID 28302699
- [Background] Luther L, Fukui S, Firmin RL, McGuire AB, White DA, Minor KS, Salyers MP. Expectancies of success as a predictor of negative symptoms reduction over 18 months in individuals with schizophrenia. Psychiatry Res. 2015 Sep 30;229(1-2):505-10. doi: 10.1016/j.psychres.2015.06.022. Epub 2015 Jun 28. PMID 26162662
- [Background] Lysaker PH, Chernov N, Moiseeva T, Sozinova M, Dmitryeva N, Alyoshin V, Faith LA, Karpenko O, Kostyuk G. Contrasting metacognitive profiles and their association with negative symptoms in groups with schizophrenia, early psychosis and depression in a Russian sample. Psychiatry Res. 2020 Sep;291:113177. doi: 10.1016/j.psychres.2020.113177. Epub 2020 Jun 7. PMID 32615314
- [Background] Lysaker PH, Gagen E, Klion R, Zalzala A, Vohs J, Faith LA, Leonhardt B, Hamm J, Hasson-Ohayon I. Metacognitive Reflection and Insight Therapy: A Recovery-Oriented Treatment Approach for Psychosis. Psychol Res Behav Manag. 2020 Apr 2;13:331-341. doi: 10.2147/PRBM.S198628. eCollection 2020. PMID 32308511
- [Background] Lysaker, P. H., & Klion, R. E. (2017). Recovery, meaning-making, and severe mental illness: A comprehensive guide to metacognitive reflection and insight therapy. Routledge.
- [Background] Lysaker PH, Kukla M, Dubreucq J, Gumley A, McLeod H, Vohs JL, Buck KD, Minor KS, Luther L, Leonhardt BL, Belanger EA, Popolo R, Dimaggio G. Metacognitive deficits predict future levels of negative symptoms in schizophrenia controlling for neurocognition, affect recognition, and self-expectation of goal attainment. Schizophr Res. 2015 Oct;168(1-2):267-72. doi: 10.1016/j.schres.2015.06.015. Epub 2015 Jul 9. PMID 26164820
- [Background] Mairs H, Lovell K, Campbell M, Keeley P. Development and pilot investigation of behavioral activation for negative symptoms. Behav Modif. 2011 Sep;35(5):486-506. doi: 10.1177/0145445511411706. Epub 2011 Jul 11. PMID 21746764
- [Background] Marcellusi A, Fabiano G, Viti R, Francesa Morel PC, Nicolo G, Siracusano A, Mennini FS. Economic burden of schizophrenia in Italy: a probabilistic cost of illness analysis. BMJ Open. 2018 Feb 8;8(2):e018359. doi: 10.1136/bmjopen-2017-018359. PMID 29439067
- [Background] Moritz S, Andreou C, Schneider BC, Wittekind CE, Menon M, Balzan RP, Woodward TS. Sowing the seeds of doubt: a narrative review on metacognitive training in schizophrenia. Clin Psychol Rev. 2014 Jun;34(4):358-66. doi: 10.1016/j.cpr.2014.04.004. Epub 2014 May 6. PMID 24866025
- [Background] Moritz S, Berna F, Jaeger S, Westermann S, Nagel M. The customer is always right? Subjective target symptoms and treatment preferences in patients with psychosis. Eur Arch Psychiatry Clin Neurosci. 2017 Jun;267(4):335-339. doi: 10.1007/s00406-016-0694-5. Epub 2016 May 18. PMID 27194554
- [Background] Moritz S, Klein JP, Lysaker PH, Mehl S. Metacognitive and cognitive-behavioral interventions for psychosis: new developments . Dialogues Clin Neurosci. 2019 Sep;21(3):309-317. doi: 10.31887/DCNS.2019.21.3/smoritz. PMID 31749655
- [Background] Moritz S, Lysaker PH. Metacognition - What did James H. Flavell really say and the implications for the conceptualization and design of metacognitive interventions. Schizophr Res. 2018 Nov;201:20-26. doi: 10.1016/j.schres.2018.06.001. Epub 2018 Jun 12. PMID 29903626
- [Background] Moritz, S., & Woodward, T. S. (2007). Metacognitive training for schizophrenia patients (MCT): a pilot study on feasibility, treatment adherence, and subjective efficacy. German Journal of Psychiatry, 10(3), 69-78.
- [Background] Philipp R, Kriston L, Lanio J, Kuhne F, Harter M, Moritz S, Meister R. Effectiveness of metacognitive interventions for mental disorders in adults-A systematic review and meta-analysis (METACOG). Clin Psychol Psychother. 2019 Mar;26(2):227-240. doi: 10.1002/cpp.2345. Epub 2018 Dec 16. PMID 30456821
- [Background] Pos K, Meijer CJ, Verkerk O, Ackema O, Krabbendam L, de Haan L. Metacognitive training in patients recovering from a first psychosis: an experience sampling study testing treatment effects. Eur Arch Psychiatry Clin Neurosci. 2018 Feb;268(1):57-64. doi: 10.1007/s00406-017-0833-7. Epub 2017 Aug 21. PMID 28828697
- [Background] Rector NA, Beck AT, Stolar N. The negative symptoms of schizophrenia: a cognitive perspective. Can J Psychiatry. 2005 Apr;50(5):247-57. doi: 10.1177/070674370505000503. PMID 15968839
- [Background] Sarkar S, Hillner K, Velligan DI. Conceptualization and treatment of negative symptoms in schizophrenia. World J Psychiatry. 2015 Dec 22;5(4):352-61. doi: 10.5498/wjp.v5.i4.352. eCollection 2015 Dec 22. PMID 26740926
- [Background] Sauve G, Lavigne KM, Pochiet G, Brodeur MB, Lepage M. Efficacy of psychological interventions targeting cognitive biases in schizophrenia: A systematic review and meta-analysis. Clin Psychol Rev. 2020 Jun;78:101854. doi: 10.1016/j.cpr.2020.101854. Epub 2020 Apr 24. PMID 32361339
- [Background] Schneider, B. C., & Andreou, C. (2014). A critical review of metacognitive training (MCT) for psychosis: Efficacy, proposed mechanisms of action and significance for functional outcomes. OA Behavioral Medicine, 1.
- [Background] Shan X, Liao R, Ou Y, Ding Y, Liu F, Chen J, Zhao J, Guo W, He Y. Metacognitive Training Modulates Default-Mode Network Homogeneity During 8-Week Olanzapine Treatment in Patients With Schizophrenia. Front Psychiatry. 2020 Mar 27;11:234. doi: 10.3389/fpsyt.2020.00234. eCollection 2020. PMID 32292360
- [Background] Strauss GP, Keller WR, Buchanan RW, Gold JM, Fischer BA, McMahon RP, Catalano LT, Culbreth AJ, Carpenter WT, Kirkpatrick B. Next-generation negative symptom assessment for clinical trials: validation of the Brief Negative Symptom Scale. Schizophr Res. 2012 Dec;142(1-3):88-92. doi: 10.1016/j.schres.2012.10.012. Epub 2012 Nov 3. PMID 23127378
- [Background] Swanson L, Griffiths H, Moritz S, Cervenka S. Metacognitive training for negative symptoms: Support for the cognitive model. Clin Psychol Psychother. 2023 Mar;30(2):486-490. doi: 10.1002/cpp.2809. Epub 2022 Dec 17. PMID 36494180
- [Background] Swanson L, Schwannauer M, Bird T, Eliasson E, Millar A, Moritz S, Griffiths H. Metacognitive training modified for negative symptoms: A feasibility study. Clin Psychol Psychother. 2022 May;29(3):1068-1079. doi: 10.1002/cpp.2692. Epub 2021 Dec 17. PMID 34792834
- [Background] Thomas EC, Luther L, Zullo L, Beck AT, Grant PM. From neurocognition to community participation in serious mental illness: the intermediary role of dysfunctional attitudes and motivation. Psychol Med. 2017 Apr;47(5):822-836. doi: 10.1017/S0033291716003019. Epub 2016 Nov 25. PMID 27884217
- [Background] Üstün, T. B., Kostanjsek, N., Chatterji, S., & Rehm, J. (Eds.). (2010). Measuring health and disability: Manual for WHO disability assessment schedule WHODAS 2.0. World Health Organization.
- [Background] Veerman SRT, Schulte PFJ, de Haan L. Treatment for Negative Symptoms in Schizophrenia: A Comprehensive Review. Drugs. 2017 Sep;77(13):1423-1459. doi: 10.1007/s40265-017-0789-y. PMID 28776162
- [Background] Velligan DI, Roberts D, Mintz J, Maples N, Li X, Medellin E, Brown M. A randomized pilot study of MOtiVation and Enhancement (MOVE) Training for negative symptoms in schizophrenia. Schizophr Res. 2015 Jul;165(2-3):175-80. doi: 10.1016/j.schres.2015.04.008. Epub 2015 May 1. PMID 25937461
- [Background] Wallwork RS, Fortgang R, Hashimoto R, Weinberger DR, Dickinson D. Searching for a consensus five-factor model of the Positive and Negative Syndrome Scale for schizophrenia. Schizophr Res. 2012 May;137(1-3):246-50. doi: 10.1016/j.schres.2012.01.031. Epub 2012 Feb 21. PMID 22356801
- [Background] Weijers, J. G., ten Kate, C., Debbané, M., Bateman, A. W., de Jong, S., Selten, J.-P. C. J., & Eurelings-Bontekoe, E. H. M. (2020). Mentalization and psychosis: A rationale for the use of mentalization theory to understand and treat non-affective psychotic disorder. Journal of Contemporary Psychotherapy: On the Cutting Edge of Modern Developments in Psychotherapy, 50(3), 223-232. doi: 10.1007/s10879-019-09449-0
- [Background] Weissman, A.; Beck, AT. Development and validation of the Dysfunctional Attitude Scale: A preliminary Investigation. Paper presented at the Education Research Association; Toronto, Ontario, Canada. 1978

DOCUMENTS (1):
  • Study Protocol (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT06127004/Prot_000.pdf